CLINICAL TRIAL: NCT05450991
Title: Long-term Qualitative and Quantitative Outcomes of Children With Hirschsprung's Disease and Anorectal Malformations
Acronym: ALOHA
Status: Recruiting | Type: Observational
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 219338
Record Dates: First submitted 2022-06-18; First posted 2022-07-11 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hirschsprung Disease; Anorectal Malformations
MeSH Terms: conditions — Hirschsprung Disease; Anorectal Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hirschsprung's Disease: Infants, children and adults cared for in Alder Hey Children's Hospital from the neonatal period onward with histologically confirmed Hirschsprung's disease.
  Interventions: Procedure: Pull through
- Anorectal Malformations: Infants, children and adults cared for in Alder Hey Children's Hospital from the neonatal period onward with an anorectal malformation.
  Interventions: Procedure: Pull through

INTERVENTIONS:
Procedure: Pull through — Children diagnosed with Hirschpsrung's Disease or an anorectal malformation, with or without operative intervention will be included
  Other Names: PSARP; Anoplasty; Soave Procedure; Swenson's Procedure; Duhammel Procedure; Cut-back

SUMMARY:
Approximately 340 babies are born with Hirschsprung's disease (HSCR) or an anorectal malformation (ARM) per year in the UK. Most require corrective surgery in the newborn or early infancy period. In both conditions, there is both variability in the severity of the condition and the type of operative technique used. Many children do well following surgery and have good continence in later life. However a significant proportion of children suffer from a lifetime of constipation or incontinence. This has a significant impact on their social and psychological welfare and is a significant burden on healthcare resources.

Due to the variation in practice, there are limited data on long-term outcomes following surgery for children with HSCR or ARMs. Where studies have been performed, they often include small numbers, non-standardised outcome measures and short follow-up periods. It is therefore difficult to ascertain the effectiveness of different management strategies. However, a recent Delphi process has been carried out to establish 10 core measures in HSCR to improve outcome reporting. This research group has a long track record in this research area, specifically in the determination of long-term outcomes of children with HSCR, leading to well cited papers within the literature. In the last 2 decades there has been a significant change in the surgical techniques used in HSCR, however the underlying evidence base for this is still lacking. This study seeks to follow-on from previous studies looking specifically at the long-term outcomes in children with HSCR. Furthermore, the aim is to widen the study to encompass all children treated at Alder Hey and also to use the same methodology to assess long-term outcomes for children with ARMs, as both groups of patients experience similar long term morbidity.

This will provide qualitative and quantitative data aiding counselling parents of children with HSCR/ARM.

DETAILED DESCRIPTION:
Hirschsprung's disease (HSCR) affects 1 in 5000 live births in the UK and is caused by a failure of development of the enteric nervous system (aganglionosis) in the distal bowel to a variable extent. Short segment HSCR, in which the aganglionic segment is restricted to the rectosigmoid region, accounts for over 80% of cases, as opposed to the more extensive long-segment HSCR which can affect the entire colon resulting in total colonic aganglionosis.

Current surgical management requires resection of the affected bowel with anastomosis of normal bowel to the anus or rectum. There are significant differences in operative and management strategies nationally and globally which include open, laparoscopic and purely trans-anal approaches, and the different pull-through procedures include the Duhamel, Swenson and the Soave. Each approach has potential advantages and disadvantages however it is not possible to draw a conclusion as to which operative strategy is the 'gold standard'.

The reasons for the current lack of clarity are multifactorial. In particular, most studies are small single-center, observational, short duration and retrospective. There is also a lack of strong evidence from systematic reviews and meta-analyses. Furthermore, there have been changes in practice over time in addition to significant outcome reporting heterogeneity in the published literature. It is therefore extremely difficult to provide accurate prognostic data to parents when the newborn is diagnosed with HSCR and at the time of the definitive pull-through procedure.

The investigators have previously reported early adult functional outcomes and long-term functional outcomes following the Duhamel procedure. Functional outcome scores were calculated by using the Rintala scoring system, and individual scores improved with time. There has since been a change in practice at Alder Hey (AH) and the more common procedure now performed is a modification of the Soave procedure. It is therefore of importance to compare the functional outcomes of patients who have undergone different procedures and to assess the longer-term outcomes of the cohort previously assessed.

Eleven years ago the investigators also published the outcomes of children with anorectal malformations (ARMs) in children presenting between 1994 and 2000. At the time the Posterior-Sagittal Ano-RectoPlasty (PSARP) had recently become the widely accepted primary surgical approach to ARMs. The study unit established a follow-up clinic dedicated solely to patients with ARM in 1994 and consultants sub-specialised to prevent dilution of case-load.

Primary outcomes were functional outcomes and quality of life. These were studied in children aged 4 years and over by the end of the study period. 85 patients qualified for the study with an age range of 4.2 to 10.1 years (median 6.7 years). 76 patients were eligible to complete the functional questionnaire and there was a response rate of 76.3% (58/76). 77.5% (62) completed the QOL score. These were compared with an age and gender-matched control group.

The study found that children with a more severe lesion had a significantly lower functional outcome score, independent of age. However, their quality of life did not seem to be impacted upon by their condition.

The long-term outcome of ARMs is poorly described. Understanding the childhood impact of ARM on a child and family's function and QOL in the medium term is important. However, the long-term impact on adolescents and adults who have this condition may differ significantly. During this period there is a significant shift in the patient's understanding and management of their own condition, and other factors including sexual function and obstetric issues become more important.

Since this study period there has been an increase in the undertaking of surgery in the neonatal period in children with a 'low' ARM, in some cases avoiding colostomy in those who would previously have required one. This change in practice may alter the impact of an ARM on a child's QOL and function.

The NETS1HD study group have recently developed a core outcome set to be used in studies comparing interventions for children with Hirschsprung's Disease which consists of a group of agreed, standardised outcomes that have been identified by key stakeholders as being the most important in determining success of treatment.

By using this core outcome set to evaluate the short and long-term outcomes of children with HSCR and ARM in the North West region, this study will be able to provide important prognostic information to parents. As this is a heterogenous group of patients, the investigators will be looking to identify the differences in long-term functional outcomes between patient subgroups and whether particular operative strategies have more favourable long-term outcomes. This will allow counselling of parents appropriately at the time of diagnosis and will assist clinical decision-making regarding the management of individual patients.

ELIGIBILITY:
Inclusion Criteria:

* All children treated at either center with histologically confirmed Hirschsprung's Disease since diagnosis from 1991
* All children diagnosed with anorectal malformation on the basis of position in relation to the external sphincter and size

Exclusion Criteria:

* Patients with non-histologically diagnosed Hirschsprung's Disease
* Patients whose initial primary treatment or majority of follow-up for either condition has been external to either center
* Patients with funnel anus
* Adults who are unable to consent for themselves

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults diagnosed with Hirschsprung's disease or Anorectal Malformation since 1991 cared for in a single centre.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Quality of life of children and adults with HSCR and ARM to pre-defined controls | 1 year of age
  PedsQL score for children. Compared to pre-defined controls. Score 0 (best)-92 (worst)
Comparison of the Quality of life of children and adults with HSCR and ARM to pre-defined controls | 5 years of age
  PedsQL score for children. Compared to pre-defined controls. Score 0 (best)-92 (worst)
Comparison of the Quality of life of children and adults with HSCR and ARM to pre-defined controls | 10 years of age
  PedsQL score for children. Compared to pre-defined controls. Score 0 (best)-92 (worst)
Comparison of the Quality of life of children and adults with HSCR and ARM to pre-defined controls | 15 years of age
  PedsQL score for children. Compared to pre-defined controls Score 0 (best)-92 (worst)
Comparison of the Quality of life of children and adults with HSCR and ARM to pre-defined controls | 20 years of age
  GI-QOL score. Compared to pre-defined controls. 0 (worst)-144 (best)
Comparison of the Quality of life of children and adults with HSCR and ARM to pre-defined controls | 30 years of age
  GI-QOL score. Compared to pre-defined controls. 0 (worst)-144 (best)
Description of urinary function of children and adults with HSCR and ARM | 5 years of age
  Proportion requiring urinary catheterisation or experiencing urinary incontinence
Description of urinary function of children and adults with HSCR and ARM | 10 years of age
  Proportion requiring urinary catheterisation or experiencing urinary incontinence
Description of urinary function of children and adults with HSCR and ARM | 15 years of age
  Proportion requiring urinary catheterisation or experiencing urinary incontinence
Description of urinary function of children and adults with HSCR and ARM | 20 years of age
  Proportion requiring urinary catheterisation or experiencing urinary incontinence
Description of urinary function of children and adults with HSCR and ARM | 30 years of age
  Proportion requiring urinary catheterisation or experiencing urinary incontinence
Comparison of the bowel function of children and adults with HSCR and ARM to pre-defined controls | 5 years 0 (worst)-52 (best)
  Paediatric incontinence and constipation score
Comparison of the bowel function of children and adults with HSCR and ARM to pre-defined controls | 10 years 0 (worst)-52 (best)
  Paediatric incontinence and constipation score
Comparison of the bowel function of children and adults with HSCR and ARM to pre-defined controls | 15 years 0 (worst)-52 (best)
  Paediatric incontinence and constipation score
Description of the Mortality rate of children and adults with ARM and HSCR | 1year of age
  Death rate with cause given
Description of the Mortality rate of children and adults with ARM and HSCR | 5 years of age
  Death rate with cause given
Description of the Mortality rate of children and adults with ARM and HSCR | 10 years of age
  Death rate with cause given
Description of the Mortality rate of children and adults with ARM and HSCR | 15 years of age
  Death rate with cause given
Description of the Mortality rate of children and adults with ARM and HSCR | 20 years of age
  Death rate with cause given
Description of the Mortality rate of children and adults with ARM and HSCR | 30 years of age
  Death rate with cause given

SECONDARY OUTCOMES:
Comparison of the sexual health of adults with HSCR and ARM compared to pre-defined controls and obstetric health | 30 years of age
  Descriptive data
Description of the obstetric health of adults with HSCR and ARM | 30 years
  Descriptive data

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No